CLINICAL TRIAL: NCT05879393
Title: The Effect of the Multistrain Probiotic OMNi-BiOTiC® Active for Upper Respiratory Tract Infections in Older People: A Randomised Controlled Trial
Brief Title: The Multistrain Probiotic OMNi-BiOTiC® Active for Upper Respiratory Tract Infections in Older People
Acronym: ProURTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Maribor (Other)
Responsible Party: Principal Investigator, Sabina Fijan, Assoc. prof. dr., University Maribor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UMaribor
Record Dates: First submitted 2023-04-27; First posted 2023-05-30 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Acute Upper Respiratory Tract Infection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multistrain Probiotic OMNi-BiOTiC® Active (Experimental): Lacticaseibacillus casei W56, Lactobacillus acidophilus W37, Ligilactobacillus salivarius W24, Levilactobacillus brevis W63, Lactococcus lactis W58, Lactococcus lactis W19, Bifidobacterium animalis subsp. lactis W52, Bifidobacterium longum subsp. longum W108, Bifidobacterium breve W25, Bifidobacterium animalis subsp. lactis W51 and Bifidobacterium bifidum W23. Additional ingredients:corn starch, maltodextrin, plant protein, potassium chloride, magnesium sulphate, manganese sulphate and vanillin
  Interventions: Dietary Supplement: OMNi-BiOTiC® Active
- Placebo (Placebo Comparator): rice starch, maltodextrin, plant protein, potassium chloride, magnesium sulphate, manganese sulphate
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: OMNi-BiOTiC® Active — Multistrain probiotic
  Arms: Multistrain Probiotic OMNi-BiOTiC® Active
Other: Placebo — rice starch, maltodextrin, plant protein, potassium chloride, magnesium sulphate, manganese sulphate
  Arms: Placebo

SUMMARY:
The goal of this randomised controlled trial is to determine the effect of consuming a multistrain probiotic OMNi-BiOTiC® Active to shorten the incidence and duration of acute upper respiratory tract infections (URTIs) in older people. The main questions it aims to answer is:

* Is the multistrain probiotic OMNi-BiOTiC® Active effective in reducing the incidence of URTIs in older people?
* Is the multistrain probiotic OMNi-BiOTiC® Active effective in reducing the duration of URTIs in older people?
* Is the multistrain probiotic OMNiBiOTiC® Active effective in changing selected immunological blood parameters in older people? Researchers will compare the probiotic group and the placebo group to see if the incidence or duration of URTIs are significant among the groups.

ELIGIBILITY:
Inclusion Criteria:

* 65 years or older at the signing of the written consent form
* ability of participant to eat independently
* ability of participant to adhere to all procedures of the clinical study

Exclusion Criteria:

* participants experienced an exacerbation of an existing chronic disease
* participants experienced an exacerbation of metabolic diseases,
* participants with mental incapacity to understand instructions
* participants were prescribed long-term usage of antibiotics.
* participants that changed their eating habits or consumed any probiotics 14 days
* participants with markedly abnormal results of blood tests were excluded.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 95 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2022-02-13 (Actual); Study Completion 2022-07-13 (Actual)

PRIMARY OUTCOMES:
Incidence of URTI | 12 weeks supplementation
  Comparison of the incidence of acute upper respiratory tract infections among older people in both arms

SECONDARY OUTCOMES:
Duration of URTI | 12 weeks supplementation
  Comparison of the duration of acute upper respiratory tract infections among older people in both arms via the use of a questionnaire
Changes in concentration of leukocytes, neutrophils segm., lymphocytes, monocytes, eosinophils, basophils in serum | 12 weeks supplementation
  Differences in the serum concentration of leukocytes, neutrophils segm., lymphocytes, monocytes, eosinophils, basophils, measured in 10x9/L of the participants in the first winter season as a change from baseline to 12 weeks upon administration of probiotics compared to placebo
Changes in concentration of Immunoglobulin A (IgA) in serum | 12 weeks supplementation
  Differences in the serum concentration of immunoglobulin A (IgA), measured in g/L of the participants in the first winter season as a change from baseline to 12 weeks upon administration of probiotics compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Sabina Fijan, Ph.D, Study Director — University of Maribor, Faculty of Health Sciences
Locations (1):
- University of Maribor, Faculty of Health Sciences, Maribor, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Strauss M, Micetic Turk D, Lorber M, Pogacar MS, Kozelj A, Tusek Bunc K, Fijan S. The Multi-Strain Probiotic OMNi-BiOTiC(R) Active Reduces the Duration of Acute Upper Respiratory Disease in Older People: A Double-Blind, Randomised, Controlled Clinical Trial. Microorganisms. 2023 Jul 5;11(7):1760. doi: 10.3390/microorganisms11071760. PMID 37512932